CLINICAL TRIAL: NCT02229981
Title: An Early-Phase Clinical Trial Evaluating ABC294640 in Patients With Refractory/Relapsed Diffuse Large B-cell Lymphoma or Kaposi Sarcoma
Brief Title: Early Phase Evaluation of ABC294640 in Patients With Refractory/Relapsed Diffuse Large B-cell Lymphoma or Kaposi Sarcoma
Acronym: ABC-102
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was discontinued due to lack of recruitment.
Sponsor: RedHill Biopharma Limited (Industry)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other); Apogee Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABC-102
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Diffuse Large B Cell Lymphoma; Kaposi Sarcoma
Keywords: Lymphoma; B-cell Lymphomas; Diffuse Large B-cell Lymphoma; Lymphosarcoma; Kaposi's Sarcoma-associated Herpesvirus; KHSV; Human Immunodeficiency Virus; HIV; Epstein-Barr Virus; EBV; Kaposi sarcoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Sarcoma, Kaposi; Lymphoma; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Acquired Immunodeficiency Syndrome; Epstein-Barr Virus Infections | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABC294640 (Experimental): Patients will receive ABC294640 orally in gelatin capsules BID.
  Interventions: Drug: ABC294640

INTERVENTIONS:
Drug: ABC294640
  Other Names: Yeliva

SUMMARY:
This is a sequential Phase I and IIa study to identify the maximum tolerated dose and to evaluate safety, tolerability, toxicity, pharmacokinetics and pharmacodynamics of the oral sphingosine kinase inhibitor ABC294640 specifically in patients with diffuse large B-cell lymphoma (DLBCL), including virus-associated (e.g., KSHV- or EBV-associated) DLBCL or Kaposi Sarcoma (KS) after failure of or intolerance to initial standard therapy.

DETAILED DESCRIPTION:
Sphingosine Kinase (SK) is an innovative target for anti-cancer therapy due to its critical role in lipid metabolism which drives cancer cell growth. We have found that the SK inhibitor ABC294640 (which is formulated for clinical use as an oral agent) significantly inhibits and reverses progression of virus-associated DLBCL in pre-clinical animal models [Qin et a., 2014]. In addition, we have found that ABC294640 selectively induces death for virus-infected endothelial cells in a laboratory model relevant to KS, with selective sparing of uninfected cells [Dai et al., 2014; Dai et al., 2015]. Both DLBCL and KS disproportionately impact patients with immune-deficiencies, including HIV infection, for whom standard chemotherapeutic approaches are less effective and incur greater side effects. Therefore, this trial which utilizes a well-tolerated, oral agent to inhibit SK for DLBCL and KS patients may provide a unique approach to treatment.

ELIGIBILITY:
Inclusion Criteria

1. Pathologically confirmed DLBCL or KS. In the case of patients with DLBCL, the disease must be radiographically refractory to standard therapy, or relapsed following standard therapy (one or more tumors measurable on PET-CT scan). In the case of patients with KS, the disease must be either radiographically or clinically refractory (persistent skin lesions) to standard therapy or relapsed following standard therapy (one or more tumors measurable on CT scan or through direct measurement of skin tumors). Please see caveats for antineoplastic therapies in Exclusion criteria below.
2. For patients with DLBCL, the patient is not a candidate for hematopoietic stem cell transplantation (as determined by medical oncologists at participating institutions) or has failed stem cell transplantation.
3. Tumor progression after receiving standard/approved chemotherapy, or lack of candidacy for standard therapy.
4. One or more tumors measurable on PET-CT scan (DLBCL), CT scan (KS), or by clinical exam of skin (KS).
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3.
6. Life expectancy of at least 3 months.
7. Age ≥ 18 years.
8. Signed, written IRB-approved informed consent.
9. A negative pregnancy test (if female).
10. Acceptable liver function:

    * Bilirubin ≤ 3 times upper limit of normal (CTCAE Grade 2 baseline)
    * AST (SGOT), ALT (SGPT) ≤ 3 x ULN (CTCAE Grade 1 baseline)
    * Serum creatinine ≤ 1.5 X ULN (CTCAE Grade 1 baseline)
11. Acceptable hematologic status:

    * Absolute neutrophil count ≥ 1000 cells/mm3
    * Platelet count ≥ 75,000 (plt/mm3) (CTCAE Grade 1 baseline)
    * Hemoglobin ≥ 8 g/dL
12. Urinalysis: No clinically significant abnormalities.
13. PT and PTT ≤ 1.5 X ULN after correction of nutritional deficiencies that may contribute to prolonged PT/PTT.
14. For men and women of child-producing potential, willingness to use of effective contraceptive methods during the study. If female (or female partner of male subject), is either not of childbearing potential (defined as postmenopausal for ≥ 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or practicing one of the following medically acceptable methods of birth control and agrees to continue with the regimen throughout the duration of the study:

    * Oral, implantable or injectable contraceptives for 3 consecutive months before the Baseline/Randomization Visit.
    * Total abstinence from sexual intercourse (≥ 1 complete menstrual cycle before the Baseline/Randomization Visit).
    * Intrauterine device (IUD).
    * Double barrier method (condoms, sponge, diaphragm or vaginal ring with spermicidal jellies or cream).

Exclusion Criteria

1. New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG.
2. Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use barrier methods (preferably condoms) or other methods of birth control at your doctor's discretion, or abstain from sexual activity, prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
3. Patients with active, life-threatening bacterial or fungal infections.
4. Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within one month prior to study entry.
5. Unwillingness or inability to comply with procedures required in this protocol.
6. Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
7. Patients who are currently receiving any other investigational agent.
8. Patients who are receiving drugs other than highly active antiretroviral therapy (HAART) or trimethoprim-sulfamethoxazole that are sensitive substrates of CYP450 1A2, 3A4, 2C9, 2D6, or 2C19, or strong inhibitors or inducers of these isozymes that cannot be stopped at least 7 days or 5 half-lives (whichever is longer) before starting treatment with ABC294640 and either replaced with another appropriate medication or not given for the duration of the clinical study. Patients on HAART will be restricted to preferred, potent agents with no demonstrated interactions with CYP450 isoforms for which significant interactions are predicted with ABC294640 (1A2, 2C9, or 2C19 for which ABC294640 IC50 < 1uM). These include tenofovir, FTC, 3TC, abacavir, darunavir, atazanavir, norvir, raltegravir, dolutegravir, elvitegravir, cobicistat, and maraviroc. Switching of ART prior to study entry is permitted given significant data for improvement/maintenance of HIV suppression when switching regimens in other contexts.
9. Patients who are currently taking Coumadin or Coumadin derivatives.
10. Patients who have received any antineoplastic therapy within 1 month of starting treatment with ABC294640 or who have not adequately recovered from side effects and toxicities of previous antineoplastic therapy.
11. Patients who are currently participating in any other clinical trial of an investigational product.
12. Allergy to radiographic contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Determine Maximum tolerated dose (MTD) of ABC294640 in patients with refractory/relapsed DLBCL or KS and determine tolerability at MTD. | Patients will be followed until a dose limiting toxicity (DLT) is experienced, if present, expected within the first 8 weeks
Evaluate safety of ABC294640 in patients with refractory/relapsed DLBCL or KS | If present, expected within 8 weeks

SECONDARY OUTCOMES:
Measure plasma levels of ABC294640 (pharmacokinetics) in patients with DLBCL or KS | Days 1 and 28, 1,2, 4, 8 and 24 hours post drug administration
Measure plasma levels of sphingosine-1-phosphate in response to ABC294640 in patients with DLBCL or KS | Days 1,8,15 and 28 in Cycle 1, Days 14 and 28 for all subsequent cycles and at the end of treatment study
Measure levels of circulating CD4+ T cell count, KSHV/EBV viral loads, and HIV viral load (if applicable) in response to ABC294640 in patients with DLBCL or KS | Days 1, 8, 15 and 22 for cycles 1-3 and Days 1, 8, 15, 22 and 28 for Cycle 4
Evaluate antitumor activity of ABC294640 in virus-associated DLBCL or KS patients by objective radiographic assessment using PET (DLBCL) or CT (KS) criteria, or measurement of clinically evident skin lesions (KS) | Within 14 Days of Treatment Day 1 and then on Day 28 of Cycles 2, 4, 6, 8, etc., stopping if tumor progression is observed

CONTACTS AND LOCATIONS:
Overall Officials: Suki Subbiah, MD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- Louisiana State University Health Sciences Center, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Qin Z, Dai L, Trillo-Tinoco J, Senkal C, Wang W, Reske T, Bonstaff K, Del Valle L, Rodriguez P, Flemington E, Voelkel-Johnson C, Smith CD, Ogretmen B, Parsons C. Targeting sphingosine kinase induces apoptosis and tumor regression for KSHV-associated primary effusion lymphoma. Mol Cancer Ther. 2014 Jan;13(1):154-64. doi: 10.1158/1535-7163.MCT-13-0466. Epub 2013 Oct 18. PMID 24140934
- [Background] Dai L, Plaisance-Bonstaff K, Voelkel-Johnson C, Smith CD, Ogretmen B, Qin Z, Parsons C. Sphingosine kinase-2 maintains viral latency and survival for KSHV-infected endothelial cells. PLoS One. 2014 Jul 10;9(7):e102314. doi: 10.1371/journal.pone.0102314. eCollection 2014. PMID 25010828
- [Background] Dai L, Trillo-Tinoco J, Bai A, Chen Y, Bielawski J, Del Valle L, Smith CD, Ochoa AC, Qin Z, Parsons C. Ceramides promote apoptosis for virus-infected lymphoma cells through induction of ceramide synthases and viral lytic gene expression. Oncotarget. 2015 Sep 15;6(27):24246-60. doi: 10.18632/oncotarget.4759. PMID 26327294